CLINICAL TRIAL: NCT03209128
Title: Savings of Hippocampus and Amygdala by Archetherapy in Cerebral Prophylactic Irradiation in Patients With Limited and / or Extended, Responsive or Stable Small Cell Lung Cancer (SCLC)
Brief Title: Cerebral Prophylactic Irradiation With Saving Hippocampus and Amygdala
Acronym: IPC
Status: Terminated | Type: Observational
Why Stopped: diffciculties to recruit patients and a lot of patients prematurely terminated
Sponsor: Centre Francois Baclesse, Luxembourg (Other)
Responsible Party: Sponsor
Other Study IDs: IPC
Record Dates: First submitted 2017-06-30; First posted 2017-07-06 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Irradiation prophyllactique cérébrale
  Interventions: Radiation: Irradiation prophyllactique cérébrale

INTERVENTIONS:
Radiation: Irradiation prophyllactique cérébrale — Irradiation prophyllactique cérébrale

SUMMARY:
Hippocampus and amygdala are parts of the brain involved in the recognition of emotions, memories, memory, language ... It is therefore very important to protect them during irradiation of the brain.

The aim of this study is to evaluate cerebral irradiation with saving hippocampus and amygdala protects these brain functions in patients with small cell lung cancer (SCLC) Radiotherapy of the brain

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Patients with a limited SCLC demonstrated histologically responsive or stable to radiochemotherapy or patients with a histologically proven extended SCLC responding to chemotherapy.
* WHO Performance Index 0-1 and / or Karnovsky Index> 70
* Possibility of long-term monitoring

Exclusion Criteria:

* Concomitant chemotherapy
* Impossibility of performing an MRI or CT without injection
* Presence of cerebral metastases
* History of cerebral irradiation at any time
* Patient suffering from severe collagenosis
* Patient with cognitive disorders with MMSE score <24

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with limited SCLC histologically proven to be responders or stable to radiochemotherapy or patients with histologically proven extended SCLC responding to chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2021-03-19 (Actual)

PRIMARY OUTCOMES:
Cognitive function | until 18 months after inclusion of patient
  Evaluate the cognitive function with Wechsler Memory Scale IV (WMS-IV) test

SECONDARY OUTCOMES:
Secondary effects according the CTCAE v.4 criteria | until 18 months after inclusion of patient
  Evaluate the toxicity according the CTCAE v.4 criteria
Appearance of brain metastases and their location | until 18 months after inclusion of patient
  Evaluate the brain control with brain MRI
Quality of life (QOL) of patients | until 18 months after inclusion of patient
  Evaluate QOL with FACT-BR test (Functional Assessment of Cancer Therapy-Brain)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Francois Baclesse, Esch-sur-Alzette, Luxembourg

IPD SHARING:
Plan to Share IPD: No